CLINICAL TRIAL: NCT04882345
Title: Evaluate the Safety and Efficacy of Almonertinib in the Treatment of Advanced NSCLC Patients With EGFR-sensitive Mutations Who Are Safety Intolerant After Osimertinib Treatment: a Prospective, Multi-center, Single-arm Clinical Trial
Brief Title: Almonertinib Treats Advanced NSCLC Patients With EGFR Mutations Who Are Safety Intolerant After Osimertinib Treatment
Acronym: ACTIVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lu Shun, Chief physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YX-L-202109
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer; EGFR Gene Mutation
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib group (Experimental): Patients meeting the criteria for inclusion and exclusion were included in the Almonertinib treatment group and received 110 mg of Almonertinib orally once a day.
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib is a class 1 new drug,the third-generation small molecule EGFR TKI, which can irreversibly and highly selectively inhibit EGFR sensitive mutations (such as exon 19 deletion and L858R mutation) and T790M resistance mutations.
  Patients meeting the criteria for inclusion and exclusion were included in the Almonertinib treatment group and received 110 mg of Almonertinib orally once a day.
  Other Names: HS-10296

SUMMARY:
This is a prospective, multi-center, single-arm clinical trial to evaluate the safety and effectiveness of Almonertinib treatment in patients with EGFR mutation positive and advanced non-small cell lung cancer (NSCLC) who are intolerant to the safety of osimertinib treatment.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical trial to evaluate the safety and effectiveness of Almonertinib treatment in patients with EGFR mutation positive and advanced non-small cell lung cancer (NSCLC) who are intolerant to the safety of osimertinib treatment. Patients meeting the criteria for inclusion and exclusion were included in the Almonertinib treatment group and received 110 mg of Almonertinib orally once a day.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old (including 18 years old) and under 75 years old (including 75 years old)
2. Histologically or cytologically diagnosed as locally advanced or metastatic NSCLC.
3. The CTCAE ≥ grade 3 AE related to osimertinib treatment in previous treatment with osimertinib, or platelet count <75×109 / L (≥CTCAE grade 2), white blood cell count <3×109 / L (≥ CTCAE grade 2), total bilirubin> 1.5×ULN (≥CTCAE grade 2), transaminase (ALT/AST)>3.0×ULN (≥CTCAE grade 2), and the toxic reaction has been alleviated or restored to ≤CTCAE grade 1 patient.
4. Tumor tissue samples diagnosed as locally advanced or metastatic NSCLC are confirmed to be EGFR sensitive mutations (including exon 19 deletion or L858R, both alone or coexist with other EGFR mutations). If the tumor tissue is accessible, it is recommended to send the tumor tissue for examination; if the tumor tissue is not accessible or the patient cannot accept a tissue biopsy, a blood sample is also acceptable.
5. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0 to 1, and it has not deteriorated in the previous 2 weeks, and the minimum expected survival is 12 weeks.
6. The patient has at least one tumor lesion that can be accurately measured at baseline, and the longest diameter at baseline is ≥10 mm (if it is a lymph node, the short diameter is required to be ≥15 mm). The selected measurement method is suitable for accurate repeat measurement, which can be computed tomography (CT) or magnetic resonance scan (MRI). If there is only one measurable lesion, it can be accepted as the target lesion, and a baseline assessment of the tumor lesion should be performed at least 14 days after the diagnostic biopsy.
7. Women of childbearing age should take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and should not breastfeed. Before starting the administration, the pregnancy test is negative, or meeting one of the following criteria proves that there is no risk of pregnancy:

   1. Postmenopausal is defined as amenorrhea for at least 12 months after the age is greater than 50 years and all exogenous hormone replacement therapy is stopped.
   2. For women younger than 50 years old, if the amenorrhea is 12 months or more after stopping all exogenous hormone treatments, and the luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels are within the laboratory postmenopausal reference value range, also It can be considered post-menopausal.
   3. Have received irreversible sterilization, including hysterectomy, bilateral ovariectomy or bilateral fallopian tube resection, except for bilateral fallopian tube ligation.
8. Male patients should use barrier contraception (i.e. condoms) from screening to 3 months after stopping the study treatment.
9. The subjects themselves participated voluntarily and signed an informed consent form in writing.

Exclusion Criteria:

1. Have received any of the following treatments:

   1. Have previously received any EGFR tyrosine kinase inhibitor treatment except osimertinib;
   2. The patient had undergone major surgery within 4 weeks before the first administration;
   3. Accept other test drugs, and within 5 half-lives;
   4. Within 7 days before the first administration of the study drug, CYP3A4 strong inhibitors, inducers, or drugs with a narrow therapeutic window that are CYP3A4 sensitive substrates have been used.
2. Patients with other malignant tumors who need standard treatment or major surgery within 2 years after the first administration of the study treatment.
3. As judged by the investigator, there are any serious or poorly controlled systemic diseases, such as poorly controlled hypertension, active bleeding-prone constitution, or active infection. No need to check for chronic diseases.
4. Refractory nausea, vomiting or chronic gastrointestinal disease, inability to swallow study drugs or having undergone extensive bowel resection may affect the full absorption of Almonertinib.
5. A history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of interstitial pneumonia requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
6. Meet any of the following cardiac examination results:

   1. The average corrected QT interval (QTc)> 470 msec obtained from 3 ECG examinations in the resting state, the Fridericia formula is used for QT interval correction (QTcF);
   2. Resting ECG suggests that there are various clinically significant rhythms, conduction or ECG morphological abnormalities (such as complete left bundle branch block, 3 degree atrioventricular block, 2 degree atrioventricular block, and PR between Period> 250 msec);
   3. There are any factors that increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death or prolonged QT of immediate family members under 40 Any concomitant drugs in the interval;
   4. Left ventricular ejection fraction (LVEF) ≤50%.
7. Insufficient bone marrow reserve or organ function, reaching the following laboratory limits:

   1. Absolute neutrophil count <1.5×109 / L;
   2. Platelet count <100×109 / L;
   3. Hemoglobin <90 g/L (<9 g/dL);
   4. Alanine aminotransferase> 2.5 times the upper limit of normal (ULN)
   5. Aspartate aminotransferase> 2.5×ULN
   6. Total bilirubin> 1.5×ULN; or Gilbert syndrome (unconjugated hyperbilirubinemia)
   7. Creatinine>1.5×ULN and creatinine clearance rate<50 mL/min (calculated by Cockcroft-Gault formula); only when creatinine>1.5×ULN, creatinine clearance rate needs to be confirmed.
8. Women who are breastfeeding or whose blood or urine pregnancy test results are positive within 3 days before the first dose of study treatment.
9. Active fungal, bacterial and/or viral infections requiring systemic treatment.
10. Have a history of hypersensitivity to any active or inactive ingredients of Almonertinib or to drugs with similar chemical structure to Almonertinib or the same class of Almonertinib.
11. Any serious or uncontrolled eye disease may increase the safety risk of the patient as judged by the doctor.
12. Patients who are judged by the investigator who may not comply well with the procedures and requirements of the study.
13. The investigator judges that there are any patients with conditions that endanger the safety of the patient or interfere with the evaluation of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of Almonertinib: Number of AEs/SAEs | Continuously throughout the study until 28 days after Termination of the treatment
  Number of adverse events (AEs)/serious adverse events (SAEs)

SECONDARY OUTCOMES:
Assess the anti-tumor activity: Progression Free Survival (PFS) | From date of baseline until the date of disease progression or discontinuation from study, assessed up to 24 months
  To assess the efficacy of Almonertinib in the treatment of advanced NSCLC patients with EGFR-sensitive mutations who are intolerant to safety after osimertinib treatment by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
Assess the anti-tumor activity: Objective response rate (ORR) | From date of baseline until the date of disease progression or discontinuation from study, assessed up to 24 months
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months.
Assess the anti-tumor activity: Disease control rate (DCR) | From date of baseline until the date of disease progression or discontinuation from study, assessed up to 24 months
  The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD assessed up to 24 months.
Assess the anti-tumor activity: Duration of response (DoR) | the time from date of documented progression or death in the absence of disease progression assessed up to 24 months.
  DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression assessed up to 24 months.
Assess the anti-tumor activity: Overall survival (OS) | an average of 4 years
  Start of study drug to Survival Endpoint through study completion, an average of 4 years.
Assess the anti-tumor activity: Depth of Remission (DepOR） | through study completion, an average of 1 year
  The depth of remission (change in tumor size) refers to the amount of change in the sum of the length of the longest diameter of the target lesion defined by RECIST 1.1 when no new lesions appear or no non-target lesions have progressed compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Li, Principal Investigator — The Affiliated Cancer Hospital of Chongqing University; Jianying Zhou, Principal Investigator — Zhejiang University; Xiuyu Cai, Principal Investigator — Sun Yat-sen University; Yueyin Pan, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China; Wenxiu Yao, Principal Investigator — Sichuan Cancer Hospital and Research Institute; Chun Huang, Principal Investigator — Tianjin Cancer Hospital; Minglei Zhuo, Principal Investigator — Peking University Cancer Hospital & Institute; Conghua Xie, Principal Investigator — Wuhan University; Meiqi Shi, Principal Investigator — Jiangsu Cancer Institute & Hospital; Qibin Song, Principal Investigator — Hubei Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No